CLINICAL TRIAL: NCT01182415
Title: Phase II Trial of Hihg-Dose Thiotepa, Busulfan, Cyclophosphamide, and Rituximab With Autologous Stem Cell Transplantation for Patients With CNS Involvement by Non-Hodgkin's Lymphoma or Primary CNS Lymphoma
Brief Title: High Dose Chemotherapy and Stem Cell Transplant for Non-Hodgkin's Lymphoma or Central Nervous System (CNS) Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Genentech, Inc. (Industry); Otsuka America Pharmaceutical (Industry); Dana-Farber Cancer Institute (Other)
Responsible Party: Principal Investigator, Yi-Bin A. Chen, MD, Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-444
Record Dates: First submitted 2010-04-30; First posted 2010-08-16 (Estimated); Results first posted 2017-12-29 (Actual); Last update posted 2023-04-06 (Actual); Status verified 2023-03

CONDITIONS: Non-Hodgkin's Lymphoma; CNS Lymphoma
Keywords: CNS involvement
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- High-dose chemotherapy with autologous stem cell transplant (Experimental)
  Interventions: Procedure: Autologous stem cell transplant; Drug: High-dose chemotherapy

INTERVENTIONS:
Procedure: Autologous stem cell transplant — Autologous stem cell transplant following high-dose chemotherapy
Drug: High-dose chemotherapy — High-dose chemotherapy with rituximab, thiotepa, busulfan, and cyclosphosphamide

SUMMARY:
Current standard treatments for lymphoma involving the central nervous system include chemotherapy or whole brain radiation therapy (WBRT). However, many patients do not respond to this treatment, and some of the patients who do respond relapse after treatment.

Previous research has shown that a stem cell transplant of a patient's own cells (autologous stem cell transplant) may be more effective for some patients with lymphoma involving the CNS. In previous research using autologous stem cell transplants for lymphoma involving the CNS, a conditioning regimen consisting of the drugs thiotepa, busulfan and cyclophosphamide (TCE) was used. These drugs have been shown to enter the nervous system.

In this research study, the investigators are adding the drug rituximab (Rituxan) to the drug cytarabine for the stem cell mobilization process. Cytarabine is a standard drug for mobilization. In addition, rituximab will be added to the conditioning regimen of thiotepa, busulfan and cyclophosphamide. Rituximab is approved by the FDA for the treatment of some types of lymphomas, but is not approved for use in lymphomas that involve the CNS. Rituximab is known to be able to enter the CNS. Previous research has suggested that it may help treat lymphoma that involves the CNS.

The goal of this research study is to see if adding rituximab to the stem cell mobilization and conditioning regimens helps treat lymphoma that involves the central nervous system.

DETAILED DESCRIPTION:
If the screening procedures confirm that you are eligible to participate in the research study you will have the following procedures.

Stem cell mobilization - this will take place over at least 9 days to prepare you to donate your stem cells for your autologous transplant. The drugs cytarabine, rituximab and Neupogen (G-CSF) will be given. You will be in the hospital for 2 days to receive the cytarabine infusions (and the 1st rituximab infusion of day 1 of stem cell mobilization). Then you will be discharged. You will receive the Neupogen injections as an outpatient.

Stem cell collection (leukapheresis) - When your doctor determines that your stem cell count is high enough you will have your stem cells collected by a procedure called leukapheresis. Leukapheresis is performed by collecting blood from a vein and processing it through a machine that removes the stem cells that are needed to produce bone marrow. The rest of the blood is returned to you through another vein. The harvested stem cells will be frozen and stored. These cells will be returned to you after you complete the conditioning regimen with high dose chemotherapy.

Conditioning regimen (high dose chemotherapy) - You will enter the hospital for the conditioning regimen and stay for about 30 days after you receive your stem cell transplant. The conditioning regimen to help kill cancer cells before your stem cell transplant will take place over 9 days. All drugs will be given intravenous (through an IV).

Infusion of stem cells (stem cell transplant) - Your cells will be given to you through your vein, similar to an IV infusion. The infusion usually takes several hours.

After you are discharged, you will be asked to return at about 4 weeks, 8 weeks, 12 weeks and 14 weeks after the stem cell transplant. At each visit you will have a physical exam, questions to measure your mental functioning, blood tests. About 14 weeks after the stem cell transplant you will have an eye exam, echocardiogram, lung function tests, whole body PET-CT scan, brain MRI or CT scan, MRI or CT of spinal cord (for patients who may have lymphoma in the spinal cord), collection of cerebral spinal fluid, and bone marrow aspiration.

You will have follow-up visits for 6 month to up to 4 years after the stem cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* One of the following clinical criteria:secondary CNS NHL; synchronous CNS NHL; relapsed PCNSL; relapsed IOL; PCNSL or IOL which has only achieved a PR after adequate initial therapy
* Must have CNS or intraocular involvement by NHL
* Subjects with secondary CNS NHL, relapsed PCNSL, or relapsed IOL will have received Salvage therapy for their CNS disease
* Subjects with synchronous CNS NHL will have received primary therapy including CNS-directed therapy
* Must demonstrate a partial or complete response of the CNS and systemic disease to pre-enrollment therapy, and must be in PR or CR at the time of enrollment
* Age >/= 18 and </= 75 years
* Life expectancy >/= 3 months
* ECOG performance status </= 2
* Must have adequate organ function as defined by the protocol

Exclusion Criteria:

* Stable or progressive CNS or systemic disease (SD orPD) at the time of enrollment
* Systemic or intrathecal chemotherapy or radiotherapy within 2 weeks prior to starting therapy on study
* Actively receiving any other study agents aimed to treat their disease
* A prior HDT-ASCT or allogeneic stem cell transplant (myeloablative or nonmyeloablative)
* Burkitt's lymphoma or acute lymphoblastic lymphoma
* A history of severe allergic reactions attributed to compounds of similar chemical or biologic composition to cytarabine, thiotepa, busulfan, cyclophosphamide, or rituximab
* Serious uncontrolled concurrent illness
* Any evidence of prior exposure to Hepatitis B virus
* HIV-positive
* Pregnant or lactating
* A history of malignancy other than NHL or PCNSL unless disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-06; Primary Completion 2015-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Bin A Chen, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

REFERENCES:
- [Result] Chen YB, Batchelor T, Li S, Hochberg E, Brezina M, Jones S, Del Rio C, Curtis M, Ballen KK, Barnes J, Chi AS, Dietrich J, Driscoll J, Gertsner ER, Hochberg F, LaCasce AS, McAfee SL, Spitzer TR, Nayak L, Armand P. Phase 2 trial of high-dose rituximab with high-dose cytarabine mobilization therapy and high-dose thiotepa, busulfan, and cyclophosphamide autologous stem cell transplantation in patients with central nervous system involvement by non-Hodgkin lymphoma. Cancer. 2015 Jan 15;121(2):226-33. doi: 10.1002/cncr.29023. Epub 2014 Sep 9. PMID 25204639

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Started | 30
Completed | 29
Not Completed | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 59 [24 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 17
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 30
Histology [Count of Participants; unit: Participants] — CLL: Chronic lymphocytic leukemia SLL: Small lymphocytic lymphoma
  Participants
    Diffuse Large B-cell Lymphoma | 27
    CLL/ SLL | 2
    Follicular Non-Hodgkin lymphoma | 1
Prior Treatment History [Count of Participants; unit: Participants]
  High-Dose Intravenous Methotrexate | 29
  High-Dose Cytarabine | 3
  Rituximab (Intravenous) | 30
  Whole brain radiation therapy (WBRT) | 2
  Other Radiation Therapy | 8

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With CNS Involvement by B-cell NHL, Relapsed PCNSL, or Relapsed PIOL Who Are Alive and Progression-free at One Year
Description: The proportion of patients with central nervous system (CNS) involvement by B-cell Non-Hodgkin's Lymphoma (NHL), relapsed primary central nervous system lymphoma (PCNSL), or relapsed primary intraocular lymphoma (PIOL) who are alive and progression-free at one year. Relapse was defined as per standard PCNSL criteria from clinical and MRI criteria.
Time Frame: 3 years
Population: The participant that was lost to follow-up was not available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Number analyzed (Participants) | 29
Participants | 28

2. Secondary Outcome: 2-year Progression Free Survival (PFS)
Description: The percentage of participants alive and without disease progression at 2 years. Disease progression was judged through clinical impression and MRI imaging.
Time Frame: 2 years
Population: The participant that was lost to follow-up was not available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Number analyzed (Participants) | 29
percentage of participants | 81 [59 to 92]

3. Secondary Outcome: 2-year Overall Survival (OS)
Description: The percentage of participants alive after two years
Time Frame: 2 years
Population: The participant that was lost to follow-up was not available for analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Number analyzed (Participants) | 29
percentage of participants | 93 [76 to 98]

4. Secondary Outcome: Response Rate
Description: The number of participants that achieved complete remission following high dose chemotherapy and autologous stem cell transplantation (ASCT). Complete remission is defined as the disappearance of all evidence of disease. Response was judged by MRI assessment.
Time Frame: 3 years
Population: The participant that was lost to follow-up was not available for analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
Number analyzed (Participants) | 29
Participants | 29

ADVERSE EVENTS:
Time Frame: From the start of treatment until disease progression, death, or until taken off study; median duration of 24 months.
Description: All grade 3 or greater adverse events were considered to be serious adverse events regardless of whether or not the adverse event was believed to be treatment related.
Arm/Group | High-dose Chemotherapy With Autologous Stem Cell Transplant
All-Cause Mortality (participants affected / at risk) | 3/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 0/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High-dose Chemotherapy With Autologous Stem Cell Transplant (N=30)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Lymphocyte count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 2 (2)
Investigations - Other, specify (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Depression (Psychiatric disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes